CLINICAL TRIAL: NCT06300463
Title: Platform Study of Immunotherapy Combinations in Colorectal Cancer Liver Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-06026214
Record Dates: First submitted 2024-02-29; First posted 2024-03-08 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer Metastatic; Liver Metastases; Colorectal Cancer
Keywords: Botensilimab; Balstilimab; Immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — balstilimab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Botensilimab and Balstilimab (Experimental): Two balstilimab infusions will be given prior to surgery and two infusions will be given after surgery, for a total of four doses. Each infusion will be scheduled approximately 3 weeks apart. On the same day as the first and third balstilimab infusions, botensilimab will also be given, for a total of two doses, one before and one after surgery.
  Interventions: Drug: Botensilimab; Drug: Balstilimab
- Botensilimab, Balstilimab, and AGEN1423 (Experimental): Two balstilimab infusions will be given prior to surgery and two infusions will be given after surgery, for a total of four doses. On the same day as each balstilimab infusion, participants will also receive AGEN1423 infusions, for a total of four doses. Each infusion will be scheduled approximately 3 weeks apart. On the same day as the first and third balstilimab + AGEN1423 infusions, botensilimab will also be given, for a total of two doses, one before and one after surgery.
  Interventions: Drug: Botensilimab; Drug: Balstilimab; Drug: AGEN1423
- Botensilimab, Balstilimab, and Radiation (Experimental): Participants will receive 3 doses of radiation prior to surgery. Additionally, two balstilimab infusions will be given prior to surgery and two infusions will be given after surgery, for a total of four doses. Each infusion will be scheduled approximately 3 weeks apart. On the same day as the first and third balstilimab infusions, botensilimab will also be given, for a total of two doses, one before and one after surgery.
  Interventions: Drug: Botensilimab; Drug: Balstilimab; Radiation: Radiation

INTERVENTIONS:
Drug: Botensilimab — 75 mg IV Q6W
  Other Names: AGEN1181
Drug: Balstilimab — 450 mg IV Q3W
  Other Names: AGEN2034
Drug: AGEN1423 — 30 mg/kg IV Q3W
  Arms: Botensilimab, Balstilimab, and AGEN1423
Radiation: Radiation — 8Gy x 3 between Day 0 - 18; Allowed techniques for radiation are 3D conformal, intensity modulated radiotherapy (IMRT), or SBRT
  Arms: Botensilimab, Balstilimab, and Radiation

SUMMARY:
The goal of this clinical trial is to to learn about different combinations of immunotherapy in patients with colorectal cancer whose cancer has spread to their liver and are planning to have surgery to remove tumor metastases from their liver. The main questions it aims to answer are:

* whether these combinations of immunotherapy change the tumor microenvironment in the liver
* whether these combinations of immunotherapy are safe and effective when used in colorectal cancer with liver metastases

Participants will be randomly assigned to one of the following:

* Botensilimab and balstilimab
* Botensilimab, balstilimab, and AGEN1423
* Botensilimab, balstilimab, and radiation

Participants will be asked to come in to receive drug infusions (and radiation, if applicable) before and after their surgical resection. Participants will be followed for up to 2 years.

DETAILED DESCRIPTION:
This is a single-center, 3-arm, randomized, open-label, phase II, screening study to assess the initial immunological changes in the tumor microenvironment in response to treatment with combination immunotherapy (Botensilimab/ Balstilimab), with or without radiation and/or additional TGFβ-CD73 trap, in patients with colorectal cancer liver metastases.

Participants who meet eligibility criteria will be randomized to receive one of 3 investigational treatment: botensilimab + balstilimab (Arm 1); botensilimab + balstilimab + AGEN1423 (Arm 2); or botensilimab + balstilimab + radiation (Arm 3). The study arms are not directly or formally compared with each other. It is established that the tumor infiltrating lymphocytes have been predictive of patient survival following resection of colorectal cancer liver metastases. Immunotherapy combinations with an increase in the ratio of CD8+ T cells: Tregs will be considered for further investigation.

All participants will have a total of four treatment visits to receive immunotherapy infusions. Two visits will occur prior to surgery, each approximately 3 weeks apart. Surgery will be scheduled between day 28-42. After surgery, you will return for two more treatment visits. After the last dose of immunotherapy, participants will come to the clinic approximately 3 weeks and 3 months later for follow-up visits. Participants will be followed remotely for up to two years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic colorectal adenocarcinoma with liver metastases
* Participant must be planning to undergo a surgical resection of their liver metastases.
* Tumor is non-MSI-H/dMMR
* Presence of measurable disease
* Participants must be willing to consent to additional molecular analyses of tumor samples removed during surgery for research purposes
* Women of childbearing potential (WOCBP), or anyone with a uterus, must not be pregnant or breastfeeding. All participants of childbearing potential must agree to use highly effective contraception during this study
* Participants may not receive chemotherapy, growth factor support, transfusions, or albumin administration within 14 days of start of study treatment.

Exclusion Criteria:

* Not eligible for surgery
* Any medical condition such as uncontrolled infection, uncontrolled diabetes mellitus or cardiac disease which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient.
* Previous allogeneic tissue/organ transplant
* Previously received PD-1, PD-L1, or CTLA-4 therapy including experimental immunologic agents
* Participants must not have any contraindications to immune checkpoint inhibitors
* Participants must not have active autoimmune disease that has required systemic treatment within 2 years prior to registration. Some exceptions are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Mean CD8:Treg ratio, as determined by flow cytometry of tumor tissue, at time of surgical resection in each treatment arm | At surgical resection
  Preliminary immunological response to treatment will be assessed by comparison of the CD8:Treg ratios in tumor tissue obtained during standard of care surgical resection between treatment arms. CD8:Treg ratio will be assessed by flow cytometry

SECONDARY OUTCOMES:
Number of Treatment-Related Adverse Events (TRAEs) as assessed by CTCAE v5.0 per treatment arm | 90 days following the last dose of study drug
  Potentially treatment-related AEs include any AEs that are assessed as possibly, probably, or definitely related to one of the study interventions. AEs will be reported by CTCAE v5.0 term.
Pathological Response Rate Per Arm | At surgical resection
  Resected tumors from the liver will be examined in their entirety, and regression of resected tumors was assessed by estimating the percentage of residual viable tumor of the macroscopically identifiable tumor bed, as identified on routine hematoxylin and eosin (H&E) staining. In addition, regression will be classified using the Mandard tumor regression grading system. Major pathologic response (MPR) will be defined as ≤10% of residual viable tumor cells (or ≥ 90% response). PR will be defined as at least 50% tumor regression. Pathological response rate will be reported as the number of patients with MPR or PR.
Radiographic Response Rate Per Arm | 90 days following the last dose of study drug
  Radiographic response will be evaluated based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Radiographic response rate will be reported as the number of patients with CR or PR.
Number of Participants Per Arm with ctDNA Clearance | 90 days following the last dose of study drug
  Circulating tumor DNA (ctDNA) will be assessed at 90 days following the last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Manish Shah, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine/NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No